CLINICAL TRIAL: NCT00845507
Title: A Double-Blind Placebo-Controlled Study of Exenatide for the Treatment of Weight Gain Associated With Olanzapine in Obese Adults With Bipolar Disorder, Major Depressive Disorder, Schizophrenia or Schizoaffective Disorder
Brief Title: Exenatide for the Treatment of Weight Gain Associated With Olanzapine in Obese Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Melissa Delbello, Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Exenatide
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Results first posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2015-08

CONDITIONS: Weight Gain
Keywords: weight gain
MeSH Terms: conditions — Weight Gain | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide Group (Experimental): Exenatide dstarted at 5 mcg subcutaneously twice daily within one hour before the morning and evening meals, and increased (as tolerated) to 10 mcg.
  Interventions: Drug: Exenatide
- Placebo Group (Placebo Comparator): Placebo: Sterile solution in equivalent doses as Exenatide
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exenatide — The dosage of study medication will be 5 mcg injection of exenatide twice daily for 28 days. On day 28 the dosage may be increased, as tolerated, to 10 mcg twice daily.
  Other Names: Exenatide (Byeta)
  Arms: Exenatide Group
Drug: Placebo — Placebo: Sterile solution in equivalent doses as Exenatide
  Arms: Placebo Group

SUMMARY:
The purpose of this research study is to test the safety and efficacy (how well it works) of exenatide as a treatment for weight gain associated with olanzapine in obese adults with Bipolar Disorder, Major Depressive Disorder, Schizophrenia or Schizoaffective Disorder

Exenatide has been approved by the FDA for the treatment of Type 2 diabetes.

It has not been approved for the treatment of weight gain associated with olanzapine in obese adults with bipolar disorder, Major Depressive Disorder, Schizophrenia or Schizoaffective Disorder

DETAILED DESCRIPTION:
Double-blind studies suggest that olanzapine is highly effective for the treatment of individuals with bipolar disorder. However, weight gain and impaired glucose tolerance remain significant concerns associated with olanzapine. Exenatide is an anti-diabetic medication that is associated with weight loss and improved glucose regulation. Therefore, the overall goal of the proposed study is to conduct a 16-week double-blind placebo-controlled study of exenatide for the treatment of weight gain associated with olanzapine in 60 obese adults with bipolar disorder treated with olanzapine. We propose to conduct the study over the course of 24 months, with an expected enrollment of approximately 3 patients per month. The primary outcome measure will be change from baseline to endpoint in weight. The secondary outcome measures will include changes from baseline to endpoint, in body mass index (BMI), abdominal circumference, metabolic parameters, clinical global improvement of psychiatric symptoms, and change in manic, depressive and psychotic symptoms. Rates of adverse events also will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be between the ages of 18 and 55 years old.
2. Subjects must have bipolar I disorder, schizophrenia, schizoaffective disorder or MDD as defined by DSM-IV-TR criteria and diagnosed using the Structured Clinical Interview for DSM-IV (SCID).
3. Subjects must have a Young Mania Rating Scale (YMRS) score < 16 and a Montgomery-Asberg Depression Rating Scale (MADRS) score < 24 at screening and baseline visits.
4. Subjects must have the Scale for the Assessment of Positive Symptoms (SAPS) scores <2 on all subscales.
5. Subjects must have gained > 7% of their body weight following treatment with olanzapine as either documented in their medical records or by patient report.
6. Subjects must be obese, as defined by a current Body Mass Index (BMI) > 30 kg/m2.
7. Subjects must sign the Informed Consent Document after the nature of the trial has been fully explained.
8. If female, subjects must be: postmenopausal, surgically incapable of childbearing, or practicing medically acceptable method(s) of contraception (e.g., hormonal methods, intrauterine device, abstinence) for at least one month prior to study entry and throughout the study.
9. Subjects must be on a stable dose of olanzapine for at least 14 days and must have been on 5-30mg/day for at least 1 month.

Major Exclusion Criteria

1. Subjects with clinically significant suicidal or homicidal ideation.
2. Subjects who have a DSM-IV lifetime diagnosis of a substance dependence disorder within the past 6 months or within the past month have been diagnosed with a substance abuse disorder, (except for nicotine abuse or dependence), as determined by psychiatric history or SCID interview.
3. Subjects with a clinically significant or unstable medical disease, including hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, immunologic, hematologic or other systemic medical conditions, that could interfere with diagnosis, assessment, or treatment of bipolar disorder or obesity, as well as subjects with a history of pancreatitis.
4. Patients with clinically significant laboratory abnormalities (> 3 times upper limit of normal), on any of the following tests: CBC with differential, electrolytes, BUN, creatinine, hepatic transaminases, lipid profile, fasting glucose, urinalysis, or thyroid indices or clinically abnormal ECG.
5. Female patients who are either pregnant or lactating.
6. Any female patient whose sexual activity is unknown or in questions.
7. Any history of current or past diabetes that has been treated with pharmacological intervention. Subjects who have a diagnosis of diabetes, are currently receiving exenatide, insulin, or an oral anti-hyperglycemic medication, or who have a nonfasting blood glucose ≥ 200 mg/dl or a fasting blood glucose ≥126 mg/dl on 2 separate tests. Subjects with pre-diabetes will not be excluded.
8. Neurological disorders including epilepsy, stroke, or severe head trauma. Mental retardation (IQ <70).

10. Treatment with an injectable depot neuroleptic within less than one dosing interval between depot neuroleptic injections and day 0.

11. Treatment with concurrent mood stabilizers (except lithium), anticonvulsants, or antipsychotics.

12. Other psychotic disorders (including delusional disorder, brief psychotic disorder, psychotic disorder due to a general medical condition, substance-induced psychotic disorder, psychotic disorder not otherwise specified) as defined in the DSM-IV.

13. Dysthymic disorder or depressive disorder not otherwise specified, bipolar disorder not otherwise specified.

14. Subjects previously enrolled in this study or have previously been treated with exenatide.

15. Subjects who have received an experimental drug within 30 days. 16. Subjects who are displaying current clinically significant depressive or manic symptoms, defined as a MADRS score >24 or a YMRS score > 16 or who currently meet DSM-IV-TR criteria for a manic, mixed, hypomanic, or depressive episode.

17. Subjects who are displaying current clinically significant psychotic symptoms, defined as any SAPS subscale score > 2 18. Subjects with a history of pancreatitis in themselves or any risk factors for developing pancreatitis (risk factors include but are not limited to: alcohol use, history of gallbladder disease or gallstones, diabetes or a family history of pancreatitis) 19. Subjects with elevated amylase or lipase levels as measured at the screening visit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2008-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa DelBello, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Patino LR, Strawn JR, Adler CM, Blom TJ, Welge JA, DelBello MP. A double-blind, placebo-controlled trial of exenatide for the treatment of olanzapine-related weight gain in obese and overweight adults. J Affect Disord. 2025 Aug 1;382:116-122. doi: 10.1016/j.jad.2025.04.046. Epub 2025 Apr 7. PMID 40203970

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Group: Placebo: Sterile solution in equivalent doses as Exenatide
  Exenatide: The dosage of study medication will be 5 mcg injection of exenatide twice daily for 28 days. On day 28 the dosage may be increased, as tolerated, to 10 mcg twice daily.
Period: Overall Study
Arm/Group | Exenatide Group | Placebo Group
Started | 24 | 30
Completed | 22 | 29
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide Group | Placebo Group | Total
Number analyzed (Participants) | 24 | 30 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (9.3) | 39.3 (11.7) | 41.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 21 | 36
  Male | 9 | 9 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 12 | 18 | 30
  Race: Non-White | 12 | 12 | 24
Region of Enrollment [Number; unit: participants]
  United States | 24 | 30 | 54
Weight [Mean (Standard Deviation); unit: Pounds] | 197 (32) | 209 (51) | 204 (44)

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight From Baseline to Endpoint.
Description: Change in weight from baseline to endpoint in the intent-to-treat (ITT) population (all subjects who took at least one dose of study medication and had one post-baseline evaluation).
Time Frame: 16 Weeks
Population: All subjects who took at least one dose of study medication and had one post-baseline evaluation.
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Exenatide Group | Placebo Group
Number analyzed (Participants) | 22 | 29
Pounds | -1.1 (6.2) | 5.9 (10.3)

2. Secondary Outcome: Change in Body Mass Index (BMI) From Baseline to Endpoint.
Description: Secondary outcome measures included change in body mass index (BMI).
Time Frame: 16 Weeks
Population: All subjects who took at least one dose of study medication and had one post-baseline evaluation.
Measure: Mean (Standard Deviation); unit: Kgs/meter squared
Arm/Group | Exenatide Group | Placebo Group
Number analyzed (Participants) | 22 | 29
Kgs/meter squared | -0.2 (1.0) | 1.0 (1.7)

ADVERSE EVENTS:
Time Frame: Up to 16 weeks
Arm/Group | Exenatide Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 2/24 | 1/30
Other Adverse Events (participants affected / at risk) | 14/24 | 11/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide Group (N=24) | Placebo Group (N=30)
Hospitalization for exacerbation of depressive symptoms (Psychiatric disorders) | 1 (1) | 1 (1)
Hospitalization for Mallory-Weiss tear (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide Group (N=24) | Placebo Group (N=30)
Gastointestinal disturbance (includes acid reflux, constipation, diarrhea, heartburn, nausea etc) (Gastrointestinal disorders) | 14 (14) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No